CLINICAL TRIAL: NCT01046916
Title: A Phase 2 Multicenter Open-label Study Evaluating the Safety and Efficacy of TAK-700 in Patients With Nonmetastatic Castration-resistant Prostate Cancer (CRPC) and a Rising Prostate-specific Antigen (PSA)
Brief Title: Safety and Efficacy Study of TAK-700 in Patients With Nonmetastatic Castration-resistant Prostate Cancer and a Rising Prostate-specific Antigen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C21001
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-700 (Experimental)
  Interventions: Drug: TAK-700

INTERVENTIONS:
Drug: TAK-700 — TAK-700 will be administered orally (PO) twice daily (BID) on a continuous schedule

SUMMARY:
This is a multicenter phase 2 open-label single-arm study that will evaluate the safety and efficacy of TAK-700 in patients with castration-resistant prostate cancer (CRPC) without radiographic evidence of metastases who have a rising prostate-specific antigen (PSA).

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria:

* Male patients 18 years or older
* Eastern Cooperative Oncology Group performance status 0-2
* Male patients who Practice effective barrier contraception during study and for 4 months after the last dose of study drug, OR Abstain from heterosexual intercourse.
* Voluntary written consent
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma without radiographic evidence of metastasis but with a rising PSA during or following the patient's most recent antineoplastic therapy despite castrate concentrations of testosterone
* Baseline PSA must be greater than or equal to 2 ng/mL and PSA doubling time must be less than or equal to 8 months OR baseline PSA must be greater than or equal to 8 ng/mL if PSA doubling time is greater than 8 months
* Has undergone orchiectomy or will continue receiving GnRH analogue therapy
* Meet screening laboratory values as specified in protocol

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Known hypersensitivity to TAK-700 or related compounds
* Received any of the following within 30 days prior to the first dose of TAK-700: any investigational compound; prior herbal product known to decrease PSA; radiation therapy for prostate cancer; OR chronic therapy with corticosteroids
* Received prior therapy with aminoglutethimide or ketoconazole
* Received antiandrogen therapy within 4 weeks for flutamide and 6 weeks for all others prior to first dose of study drug
* Received prior chemotherapy for prostate cancer
* Current bladder neck outlet obstruction caused by prostate cancer, current spinal cord compression, or current bilateral hydronephrosis
* Symptoms that investigator deems related to prostate cancer
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* History of adrenal insufficiency
* Uncontrolled cardiovascular condition
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Unwilling or unable to comply with protocol
* Major surgery or serious infection within 14 days of first dose of TAK-700
* Life-threatening illness unrelated to cancer
* Uncontrolled nausea, vomiting or diarrhea
* Known gastrointestinal disease or procedure that could interfere with oral absorption or tolerance of TAK-700

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the percentage of patients who achieve a PSA less than or equal to 0.2 ng/mL following 3 months of TAK-700 treatment | 3 months

SECONDARY OUTCOMES:
To determine PSA response rate (PSA decline of at least 90%, 50% and 30% from baseline)at 3 and 6 months | 3 and 6 months
To determine the percentage of patients who achieve a PSA less than or equal to 0.2 ng/mL following 6 months of TAK-700 treatment | 6 months
To determine time to PSA progression, time to metastases, and duration of progression-free survival | Evidence of PSA or disease progression
To monitor changes in endocrine markers | Evidence of PSA or disease progression
To evaluate the safety of TAK-700 | Evidence of PSA or disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Hussain M, Corn PG, Michaelson MD, Hammers HJ, Alumkal JJ, Ryan CJ, Bruce JY, Moran S, Lee SY, Lin HM, George DJ; Prostate Cancer Clinical Trials Consortium, a program of the Department of Defense Prostate Cancer Research Program and the Prostate Cancer Foundation. Phase II study of single-agent orteronel (TAK-700) in patients with nonmetastatic castration-resistant prostate cancer and rising prostate-specific antigen. Clin Cancer Res. 2014 Aug 15;20(16):4218-27. doi: 10.1158/1078-0432.CCR-14-0356. Epub 2014 Jun 25. PMID 24965748